CLINICAL TRIAL: NCT07277309
Title: Promoting Recovery After Brain Injury Using Focused Ultrasound
Acronym: ReBOUND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michael J. Young, M.D., M.Phil, PI, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P002816; 1K23NS140495 (NIH)
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Consciousness Disorders; Disorders of Consciousness Due to Severe Brain Injury
Keywords: Disorder of Consciousness; Vegetative State; Minimally Conscious State; Minimally Conscious State Plus; Minimally Conscious State Minus; Traumatic Brain Injury; CVA (Cerebrovascular Accident); Anoxia, Brain; Thalamic Infarction; Coma; Prolonged
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State; Brain Injuries, Traumatic; Stroke; Hypoxia, Brain; Coma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- LIFUP group (Experimental): Participants will receive low-intensity focused ultrasound intervention. Participants are also anticipated to undergo advanced MRI and EEG. Surrogate decision makers (family members) and recovered patients will undergo a semi-structured interview.
  Interventions: Device: Low-intensity focused ultrasound

INTERVENTIONS:
Device: Low-intensity focused ultrasound — Low-intensity focused ultrasound pulsations (LIFUP) will be delivered to the brain, along with advanced MRI and EEG. Surrogate decision makers (family members) and recovered patients will undergo a semi-structured interview.

SUMMARY:
The overall aim of this study is to develop an intervention that can help recovery in patients surviving severe brain injury but failing to fully recover. In particular, this project aims to (1) determine neurobehavioral responses to low-intensity focused ultrasound (LIFUP) in patients with disorders of consciousness (DoC) following brain injury, (2) determine neurophysiologic (EEG) responses to LIFUP in patients with DoC and (3) identify and evaluate ethical perspectives of patient representatives (family members and surrogate decision-makers) surrounding investigation of therapeutic neuromodulation technologies such as LIFUP in patients with DoC.

DETAILED DESCRIPTION:
Aim 1: Determine neurobehavioral responses to LIFUP in patients with DoC. Aim 2: Determine neurophysiologic (EEG) responses to LIFUP in patients with DoC.

Aim 3: Identify and evaluate ethical perspectives of patient representatives (family members and surrogate decision-makers) surrounding investigation of therapeutic neuromodulation technologies such as LIFUP in patients with DoC.

Advanced MRI will be obtained to determine predictive neuroimaging signatures of responsiveness. This project will crucially inform the groundwork for a personalized, connectome-based approach to impactful therapeutic intervention for patients affected by DoC due to diverse pathologies across the brain injury care continuum and will inform an ethical framework for responsible development and deployment of therapeutic neuromodulation technologies.

ELIGIBILITY:
Inclusion Criteria:

* Brain injury resulting in DoC diagnosis, following international guidelines
* At least 18 years of age
* Legally authorized representative (surrogate) available to consent

Exclusion Criteria:

* History of neurological disorder other than the brain injury
* Metal implant or other condition precluding MRI
* Manifest continuous spontaneous movement (which would prevent safe/successful MRI)
* Participation in concurrent therapeutic study
* Pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Determine neurobehavioral responses to LIFUP in patients with DoC: Coma Recovery Scale - Revised (CRS-R) | Days 1-3
  Outcome measures collected prior to LIFUP sessions will be compared to outcome measures obtained after LIFUP sessions. The Coma Recovery Scale Revised (CRS-R) ranges from 0 to 23 points, with higher scores indicating better neurobehavioral function and level of consciousness. The CRS-R consists of 6 subscales designed to assess auditory function, receptive and expressive language, visuoperception, communication ability, motor functions, and arousal level. The lowest score on each sub-scale represents reflexive activity; the highest represents behaviors mediated by cognitive input. The total score ranges between 0 (worst) and 23 (best).
Determine neurobehavioral responses to LIFUP in patients with DoC: Disability Rating Scale (DRS) | Days 1-3
  Outcome measures collected prior to LIFUP sessions will be compared to outcome measures obtained after LIFUP sessions. The DRS ranges from 0 to 30 points, with higher scores indicating more severe disability. DRS subscale scores include eye opening [score range 0-3], communication [score range 0-4], motor response [score range 0-5], cognitive ability for feeding [score range 0-3], cognitive ability for toileting [score range 0-3], cognitive ability for grooming [score range 0-3], level of function [score range 0-5], and employability [score range 0-3]. Subscale scores are summed to produce the total score.
Determine neurophysiologic responses to LIFUP in patients with DoC | Days 1-3
  Using electroencephalography (EEG) recordings, we will compute power spectral density within predefined frequency bands and derive ABCD-level classifications, resting-state complexity metrics, and responsiveness indices that quantify the degree of thalamocortical disconnection.
Identify and evaluate ethical perspectives of patient representatives surrounding investigation of therapeutic neuromodulation technologies such as LIFUP in patients with DoC | Days 1-3
  Family members or surrogate decision-makers (i.e., legally authorized healthcare proxies of study participants with DoC), will be engaged in interviews to capture their expectations, perspectives, and concerns surrounding the use and deployment of neuromodulation techniques in the context of brain injury. The semi-structured interview will center on key themes: hopes and expectations for neuromodulation technology; views on the informed consent process and data privacy related to neural data; considerations of equity in access to neuromodulation therapies; areas of uncertainty or concern regarding risks and benefits; and perceived roles of caregivers and families in the neuromodulation decision-making process. This approach is designed to elicit a nuanced understanding of ethical considerations as viewed by those most impacted, thereby informing a robust ethical framework that aligns research and clinical practices with the values and needs of patients and their families.

SECONDARY OUTCOMES:
Brain MRI-derived responsiveness index (structural-functional signature predicting LIFUP response) | Day 1
  Participants who can safely undergo MRI will receive an advanced brain imaging protocol. The primary quantitative measure will be a composite Brain MRI-derived Responsiveness Index, computed from predefined brain MRI features. Structural and functional metrics will be combined into a single composite index using a prespecified analytic model. The composite index will be reported as a unitless continuous score, with higher values corresponding to imaging patterns associated with greater likelihood of LIFUP responsiveness.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital (The General Hospital Corp.), Boston, Massachusetts
  - Spaulding Rehabilitation Hospital Corporation, Inc., Cambridge, Massachusetts